CLINICAL TRIAL: NCT06951516
Title: How Single-Word and Telegraphic Simplification Affects Language Processing and Word Learning in Young Children With Down Syndrome
Brief Title: How Simplified Language Affects Comprehension and Learning in Young Children With Down Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Courtney E. Venker, Associate Professor, Michigan State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3R01DC020165-02S1 (NIH)
Record Dates: First submitted 2025-04-16; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Down Syndrome
Keywords: Down syndrome; language development; language processing; language input
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Utterance Type (Experimental): This study uses a within-participant experimental manipulation. All participants will be exposed to all utterances types (across trials).
  Interventions: Behavioral: Linguistic simplification

INTERVENTIONS:
Behavioral: Linguistic simplification — Children will participate in screen-based language processing and word learning tasks in which they hear utterances with different types and amounts of linguistic simplification (i.e., a within-group manipulation).

SUMMARY:
The long-term study goal is to experimentally evaluate the components (and likely active ingredients) of early language interventions for young children with Down syndrome (DS). The overall objective is to determine how single-word and telegraphic simplification affects real-time language processing and word learning in young children with DS (relative to full, grammatical utterances). The proposed project will investigate three specific aims: 1) Determine how single-word and telegraphic simplification affects language processing. 2) Determine how single-word and telegraphic simplification affects word learning. 3) Evaluate child characteristics that may moderate the effects of linguistic simplification on language processing and word learning. Aim 1 will test the hypothesis that children with DS will process grammatical utterances faster and more accurately than telegraphic or single-word utterances. Aim 2 will test the hypothesis that overall, children will demonstrate better word learning in the grammatical compared to the single-word and telegraphic conditions. Aim 3 will test the hypothesis that receptive language and nonverbal cognitive abilities will be significant moderators, such that children with stronger linguistic and cognitive skills will show the greatest benefit from grammatical input but children with lower linguistic and cognitive scores will perform similarly across conditions.

ELIGIBILITY:
Inclusion Criteria:

* Down syndrome

English as primary language

2-7 years old

Exclusion Criteria:

* Acquired brain injury

Cerebral palsy

Uncorrected vision or hearing impairment

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Gaze location on Looking-While-Listening (LWL) tasks | Baseline
  LWL involves a child looking at a screen with two images, one on each side of the screen, while being provided an auditory cue that includes the name of the target image. The primary outcome is a dichotomous variable indicating whether the child is fixated on the target image or the distracter image; gaze directed at neither image will be considered missing. It will be determined whether gaze is to the left or right image, using trained coders who are blind to target side. Gaze location will be observed every 33 ms from 300 ms after onset to 2000 ms after target word onset, for a total of 51 observations per trial. Analyses will focus on differences across trial types and child characteristics in the trajectory of gaze location over the course of the trial.

SECONDARY OUTCOMES:
Gaze location in Teaching Phase of Study 2b (Fast Mapping) | Baseline
  A secondary outcome measure will be gaze location during the Teaching Phase of the Fast Mapping task (Study 2b). The variable is a dichotomous variable indicating whether the child is fixated on the novel image (only a single image is presented in each trial during the Teaching Phase) or not. It will be determined whether gaze is directed to the novel image, as our prior attempts to manually code single-object trials have not been successful. Only children who successfully calibrate and provide adequate automatic eye-tracking data in the Fast Mapping task will be included. Gaze location will be observed every 33 ms during the Teaching Trials. Analyses will focus on differences across trial types (single-word vs. full, grammatical teaching utterances).

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Venker, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States